CLINICAL TRIAL: NCT02642497
Title: Efficacy of Postoperative Analgesia Offered by Local Ketamine Wound Instillation Following Total Thyroidctomy; a Randomized, Double-blind, Controlled-clinical Trial
Brief Title: Local Ketamine Instillation for Postoperative Analgesia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmad Mohammad Abd El-Rahman, lecturer of anesthesia, ICU, and pain management, Assiut University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 342
Record Dates: First submitted 2015-12-24; First posted 2015-12-30 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Postoperative Pain
Keywords: postoperative analgesia; ketamine; total thyroidectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- local ketamine group (Active Comparator): intra-wound instillation of ketamine (1 mg/ kg) and normal saline in a total volume of 10 ml dispersed evenly throughout the wound; given after hemostasis and before wound closure, with closure of suction drain tube for 30 min. postoperatively.
  Interventions: Drug: intra-wound instillation of ketamine
- control group (Placebo Comparator): intra-wound instillation of normal saline in a total volume of 10 ml dispersed evenly throughout the wound; given after hemostasis and before wound closure, with closure of suction drain tube for 30 min. postoperatively.
  Interventions: Drug: intra-wound instillation of normal saline
- systemic ketamine group (Active Comparator): Intra-muscular injection of ketamine at a dose of 1 mg/kg before wound closure.
  Interventions: Drug: systemic administration of ketamine

INTERVENTIONS:
Drug: intra-wound instillation of ketamine — intra-wound instillation of ketamine (1 mg/ kg) and normal saline in a total volume of 10 ml dispersed evenly throughout the wound; given after hemostasis and before wound closure
  Arms: local ketamine group
Drug: intra-wound instillation of normal saline — intra-wound instillation of normal saline in a total volume of 10 ml dispersed evenly throughout the wound; given after hemostasis and before wound closure
  Other Names: placebo
  Arms: control group
Drug: systemic administration of ketamine — intra-muscular administration of ketamine (1 mg/ kg), given before wound closure.
  Arms: systemic ketamine group

SUMMARY:
This study aims at exploring the analgesic efficacy, and safety of Ketamine instillation into the wound of total thyroidectomy compared to placebo,and to systemic ketamine administration (I.M. injection of the same dose) with respect to postoperative VAS, first request of analgesia, total opioid consumption, and with respect to possible side effects.

ELIGIBILITY:
Inclusion Criteria:

* patients with thyroid cancer scheduled for total thyroidectomy.

Exclusion Criteria:

1. BMI>35
2. Unstable ischaemic cardiac disease
3. Increased intracranial pressure
4. Increased intraocular pressure
5. Hypersensitivity or allergy to ketamine, local anesthetic, morphine, or other drugs used in the study.
6. Severe psychiatric disease
7. Unwillingness or inability to use PCA-device
8. Inability to use VAS scale

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2015-08; Primary Completion 2016-02 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
total opioid consumption | 24 hours
  the total amount of morphine consumed during follow up period

SECONDARY OUTCOMES:
first request of analgesia | 24 hours
  time to first request of rescue analgesic drug
VAS | 24 hours
  effect of study drugs on postoperative pain measured by VAS score

OTHER OUTCOMES:
possible side effects | 24 hours
  occurrence of possible side effects during follow up

IPD SHARING:
Plan to Share IPD: Undecided